CLINICAL TRIAL: NCT01190124
Title: Raltegravir With Optimized Background Therapy (OBT) in Multiple Experienced HIV-infected Patients: a Retrospective Analysis of a Portuguese Cohort Treated Within the Expanded Access Program
Brief Title: Raltegravir With Optimized Background Therapy (OBT) in Multiple Experienced HIV-infected Patients
Status: Completed | Type: Observational
Sponsor: Doroana, Maria Manuela, M.D. (Individual)
Collaborators: Merck Sharp & Dohme LLC (Industry); Eurotrials Brasil Consultores Cientificos Ltda (Industry)
Responsible Party: Maria Manuela Doroana, MD, Hospital de Santa Maria - Centro Hospitalar Lisboa Norte
Other Study IDs: CohortHIV2008PT
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: HIV infections; HIV-1; HIV-2; Acquired Immunodeficiency Syndrome; AIDS; Anti-Retroviral Agents; Raltegravir; Integrase Inhibitors; multiple-experienced HIV infected patients
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CohortHIV: Adult multiple-experienced HIV infected patients who needed to change their antiretroviral therapy and initiated raltegravir + optimized background therapy under the Early Access Program.

SUMMARY:
The purpose of this study is to evaluate the efficacy of raltegravir with optimized background therapy (OBT) in multiple-experienced HIV infected patients, measured by the proportion of patients with undetectable viral load and the mean increase of CD4 cells count at week 24 and 48.

It is also intended to evaluate:

* viral load suppression and the mean increase of CD4 cells count at week 24 and 48 in patients who needed to change antiretroviral (ARV) therapy due to inacceptable toxicity, as determined by the investigator, including patients who needed to replace T20.
* efficacy of raltegravir with OBT in HIV-2 infected patients that were included in this cohort, measured by the percentage of patients with undetectable viral load and the mean change of CD4 cells count at week 24 and 48.

Study hypotheses:

* Raltegravir with OBT is effective in achieving and maintaining a long term virologic suppression along with a significant increase on CD4 cells count in both HIV-1 and HIV-2 infected patients.
* Patients who replaced T20 by raltegravir, due to intolerance, are able to maintain long term virologic suppression.

DETAILED DESCRIPTION:
Considering its novel mechanism of action, potency, safety and tolerability, and pharmacokinetic profile, raltegravir has been used in several clinical scenarios. Since its initial clinical use in multiresistant patients throughout the Expanded Access and Compassionate Use Program (started in March 2007) raltegravir has been used successfully in other clinical scenarios, including but not limited to: enfuvirtide-related serious adverse events and intolerance, nucleoside analogue inhibitors' toxicity, ritonavir and protease inhibitor intolerance and to avoid significant drug-drug interactions. Early access to raltegravir was basically focused on patients on therapeutic failure and triple-class resistance and due to enfuvirtide intolerance. In order to achieve a better understanding of the efficacy and safety profile of raltegravir in the clinical setting, it is intended to evaluate retrospectively HIV patients treated in Portugal with raltegravir since the Early Access and Compassionate Use Program (EAP) was implemented.

This is a national, multicenter, observational, clinical cohort study with retrospective collection of data. Each site will include patients who had started treatment with raltegravir under the EAP.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 18 years or older
2. ARV multi-experienced patients (i.e. experienced at least two prior regimens) with need to change current ARV therapy, including:

   * HIV-1 infected patients with documented therapeutic failure,
   * HIV-2 infected patients with documented therapeutic failure
   * HIV infected patients in virologic suppression who needed to change ARV due to inacceptable toxicity, as determined by the investigator, including patients who needed to replace T20
3. Raltegravir-naïve patients who initiated raltegravir since the EAP Program, with optimized background therapy(OBT)
4. Patient who has been followed at the same clinical site since the start of raltegravir

Exclusion Criteria:

1. Acute or decompensated chronic hepatitis. Patients with serum aminotransferase levels 10 times the upper limit of the normal range or higher (grade 4)
2. Patients who presented resistance to drugs included in OBT (namely, etravirine, darunavir or maraviroc)
3. Non-existing medical records for viral load and TCD4 at baseline, week 24 and 48

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected adult portuguese patients who started treatment with raltegravir since the Early Access Program and Compassionate Use Program (from March 2007 to December 2008)
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuela S Doroana, MD, Principal Investigator — Hospital de Santa Maria - Centro Hospitalar Lisboa Norte

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective collection of data took place in 11 portuguese public hospitals. Each site included patients who started treatment with raltegravir from March 2007 until December 2008.
Pre-assignment Details: 197 patients were included in the database. However, only 151 patients were included in the analysis, as 46 did not meet inclusion/exclusion criteria
Groups:
- HIV-1 at Virologic Failure: Adult multiple-experienced HIV-1 infected patients at virologic failure (patients under treatment with RNA HIV >1000 cop/mL)
- HIV With Need for Therapy Change: Adult HIV infected patients at virologic suppression (with RNA HIV <40 cop/mL), who needed to change antiretroviral therapy due to inacceptable toxicity, as determined by the investigator (including patients who needed to replace T20)
- HIV-2 With Therapeutic Failure: Adult HIV-2 infected patients with therapeutic failure (including those at virologic suppression but with decreasing immunological response with prior treatment)
Period: Overall Study
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure
Started | 107 | 24 | 20
Completed | 90 | 24 | 19
Not Completed | 17 | 0 | 1
Not completed — Death | 3 | 0 | 0
Not completed — Therapeutic Failure | 12 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure | Total
Number analyzed (Participants) | 107 | 24 | 20 | 151
Age Continuous [Median (Full Range); unit: years] | 44.0 (10.2) [30 to 77] | 45.5 (12.7) [25 to 72] | 52.5 (11.6) [27 to 65] | 45.0 (10.9) [25 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 5 | 10 | 37
  Male | 85 | 19 | 10 | 114

OUTCOME MEASURES:

1. Primary Outcome: HIV-RNA Levels
Description: Patients with undetectable viral load (confirmed HIV RNA < 50 copies/mL) at baseline.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 107 | 24 | 20
participants
  < 50 copies/mL | 0 | 24 | 10
  >= 50 copies/mL | 107 | 0 | 10
Statistical Analysis 1: Comparison: HIV-1 at Virologic Failure vs HIV With Need for Therapy Change vs HIV-2 With Therapeutic Failure; Comparison between the 3 study groups, in order to determine if there are statistically significant differences concerning HIV-RNA levels at baseline; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Primary Outcome: HIV-RNA Levels
Description: Patients achieving undetectable viral load (confirmed HIV RNA < 50 copies/mL) at week 24.
Time Frame: week 24
Measure: Number; unit: participants
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 107 | 24 | 20
participants
  < 50 copies / mL | 75 | 24 | 17
  >= 50 copies / mL | 27 | 0 | 2
  Missing value | 5 | 0 | 1

3. Primary Outcome: HIV-RNA Levels
Description: Patients achieving undetectable viral load (confirmed HIV RNA < 50 copies/mL) at week 48.
Time Frame: week 48
Measure: Number; unit: participants
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 107 | 24 | 20
participants
  < 50 copies/mL | 74 | 24 | 16
  >= 50 copies/mL | 18 | 0 | 3
  Missing value | 15 | 0 | 1

4. Primary Outcome: CD4 Cells Count
Description: CD4 cells count at baseline.
Time Frame: Baseline
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 107 | 24 | 20
cells/mm^3 | 166.00 (203.57) [3 to 856] | 391 (200.77) [120 to 925] | 120 (104.66) [15 to 430]
Statistical Analysis 1: Comparison: HIV-1 at Virologic Failure vs HIV With Need for Therapy Change vs HIV-2 With Therapeutic Failure; Comparison between the 3 study groups, in order to determine if there are statistically significant differences concerning CD4 cells count at baseline; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

5. Secondary Outcome: HIV-RNA Levels
Description: For patients in whom T20 was replaced by raltegravir it will be determined the number of patients that presented undetectable viral load (confirmed HIV RNA < 50 copies/mL) at baseline.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- HIV Patients With Therapy Replacement: HIV infected patients in whom T20 was replaced by raltegravir
Arm/Group | HIV Patients With Therapy Replacement
Number analyzed (Participants) | 20
participants
  < 50 copies/mL | 20
  >= 50 copies/mL | 0

6. Secondary Outcome: HIV-RNA Levels
Description: For patients in whom T20 was replaced by raltegravir it will be determined the number of patients that maintain undetectable viral load (confirmed HIV RNA < 50 copies/mL) at week 24.
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | HIV Patients With Therapy Replacement
Number analyzed (Participants) | 20
participants
  < 50 copies/mL | 20
  >= 50 copies/mL | 0

7. Secondary Outcome: HIV-RNA Levels
Description: For patients in whom T20 was replaced by raltegravir it will be determined the number of patients that maintain undetectable viral load (confirmed HIV RNA < 50 copies/mL) at week 48.
Time Frame: Week 48
Measure: Number; unit: participants
Arm/Group | HIV Patients With Therapy Replacement
Number analyzed (Participants) | 20
participants
  < 50 copies/mL | 20
  >= 50 copies/mL | 0

8. Secondary Outcome: CD4 Cells Count
Description: For patients in whom T20 was replaced by raltegravir CD4 cells count will be assessed.
Time Frame: Baseline
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | HIV Patients With Therapy Replacement
Number analyzed (Participants) | 20
cells/mm^3 | 400.50 (193.50) [120 to 925]

9. Secondary Outcome: CD4 Cells Count
Description: For patients in whom T20 was replaced by raltegravir it will be assessed the median changes of CD4 cells count at week 24.
Time Frame: Week 24
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | HIV Patients With Therapy Replacement
Number analyzed (Participants) | 20
cells/mm^3 | 378.00 (171.00) [171 to 864]

10. Secondary Outcome: CD4 Cells Count
Description: For patients in whom T20 was replaced by raltegravir it will be assessed the median changes of CD4 cells count at week 48.
Time Frame: Week 48
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | HIV Patients With Therapy Replacement
Number analyzed (Participants) | 107
cells/mm^3 | 452.00 (181.99) [170 to 823]

11. Secondary Outcome: CD4 Cells Count
Description: For the HIV-2 infected patients CD4 cells count will be assessed at baseline.
Time Frame: Baseline
Measure: Median (Full Range); unit: cells/mm^3
Groups:
- HIV-2 With Therapeutic Failure: Adult HIV-2 infected patients with therapeutic failure
Arm/Group | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 20
cells/mm^3 | 120.00 (104.66) [15 to 430]

12. Secondary Outcome: CD4 Cells Count
Description: For the HIV-2 infected patients CD4 cells count will be assessed at week 24.
Time Frame: Week 24
Description (as registered): For patients in whom T20 was replaced by raltegravir it will be assessed the median changes of CD4 cells count at week 24.
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 20
cells/mm^3 | 190.00 (156.83) [57 to 591]

13. Secondary Outcome: CD4 Cells Count
Description: For the HIV-2 infected patients CD4 cells count will be assessed at week 48.
Time Frame: Week 48
Description (as registered): For patients in whom T20 was replaced by raltegravir it will be assessed the median changes of CD4 cells count at week 48.
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 20
cells/mm^3 | 180.00 (160.00) [49 to 703]

14. Secondary Outcome: HIV-RNA Levels
Description: For the HIV-2 infected patients it will be determined the number of patients with undetectable viral load (confirmed HIV RNA < 50 copies/mL) at baseline.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 20
participants
  < 50 copies/mL | 10
  >= 50 copies/mL | 10

15. Secondary Outcome: HIV-RNA Levels
Description: For the HIV-2 infected patients it will be determined the number of patients that achieve or maintain undetectable viral load (confirmed HIV RNA < 50 copies/mL) at week 24.
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 20
participants
  < 50 copies/mL | 17
  >= 50 copies/mL | 2
  Missing value | 1

16. Secondary Outcome: HIV-RNA Levels
Description: For the HIV-2 infected patients it will be determined the number of patients that achieve or maintain undetectable viral load (confirmed HIV RNA < 50 copies/mL) at week 48.
Time Frame: Week 48
Measure: Number; unit: participants
Arm/Group | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 20
participants
  < 50 copies/mL | 16
  >= 50 copies/mL | 3
  Missing value | 1

17. Primary Outcome: CD4 Cells Count
Description: CD4 cells count at week 24.
Time Frame: week 24
Description (as registered): For the HIV-2 infected patients CD4 cells count will be assessed at week 24.
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 107 | 24 | 20
cells/mm^3 | 299.50 (272.28) [26 to 1409] | 389.00 (183.18) [171 to 864] | 190.00 (156.83) [57 to 591]
Statistical Analysis 1: Comparison: HIV-1 at Virologic Failure vs HIV With Need for Therapy Change vs HIV-2 With Therapeutic Failure; Comparison between the 3 study groups, in order to determine if there are statistically significant differences concerning CD4 cells count at week 24; Test type: Superiority or Other; p = 0.007, Kruskal-Wallis

18. Primary Outcome: CD4 Cells Count
Description: CD4 cells count at week 48.
Time Frame: week 48
Description (as registered): For the HIV-2 infected patients CD4 cells count will be assessed at week 48.
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure
Number analyzed (Participants) | 107 | 24 | 20
cells/mm^3 | 336.50 (3108.80) [18 to 29760] | 452.00 (174.25) [170 to 823] | 180.00 (160.26) [49 to 703]
Statistical Analysis 1: Comparison: HIV-1 at Virologic Failure vs HIV With Need for Therapy Change vs HIV-2 With Therapeutic Failure; Comparison between the 3 study groups, in order to determine if there are statistically significant differences concerning CD4 cells count at week 48; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis

19. Secondary Outcome: Adverse Drug Reactions
Description: Number of participants that suffered clinical and laboratory-associated adverse events, including events that lead to discontinuations or death. Investigator will collect all drug-related adverse events, i.e. judged by the investigator to be definitely, probably, or possibly related to the study drug.
Time Frame: Week 48
Measure: Number; unit: participants
Groups:
- Total: Total number of patients studied
Arm/Group | Total
Number analyzed (Participants) | 151
participants
  At least one adverse reaction | 12
  At least one non serious adverse reaction | 9
  At least one serious adverse reaction | 3
  Patients that discontinued due to adverse reaction | 0

ADVERSE EVENTS:
Arm/Group | HIV-1 at Virologic Failure | HIV With Need for Therapy Change | HIV-2 With Therapeutic Failure
Serious Adverse Events (participants affected / at risk) | 3/107 | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 7/107 | 1/24 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-1 at Virologic Failure (N=107) | HIV With Need for Therapy Change (N=24) | HIV-2 With Therapeutic Failure (N=20)
Edema of the lower extremities (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Toxidermia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-1 at Virologic Failure (N=107) | HIV With Need for Therapy Change (N=24) | HIV-2 With Therapeutic Failure (N=20)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated CPK (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Elevated AST/ALT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No